CLINICAL TRIAL: NCT03607175
Title: Randomized Clinical Control Trial Comparing the Effects of a Steroid Eluting Implant Versus Triamcinolone-impregnated Carboxymethylcellulose Foam on the Postoperative Clinic Experience in Patients That Underwent Functional Endoscopic Surgery for Nasal Polyposis
Brief Title: Adjunctive Treatment for Chronic Rhinosinusitis With Nasal Polyposis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marina Boruk (Other)
Collaborators: State University of New York - Downstate Medical Center (Other)
Responsible Party: Sponsor-Investigator, Marina Boruk, Principal Investigator, State University of New York - Downstate Medical Center
Organization: State University of New York - Downstate Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1161972-3
Record Dates: First submitted 2018-07-23; First posted 2018-07-31 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Chronic Rhinosinusitis; Nasal Polyps
MeSH Terms: conditions — Nasal Polyps | interventions — Triamcinolone

STUDY DESIGN:
Intervention Model Description: Study is an intrapatient control design, each subject will receive both interventions, one in each nostril
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcomes assessor will be blinded to the side that the steroid eluting implant and the triamcinolone-impregnated foam in on.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Steroid-eluting implant (Propel) (Active Comparator): Mometasone furoate implant. 370ug of mometasone furoate with each application. One application to be used at the conclusion of surgery and left in place for 1 month or less depending on if it requires removal during office debridement.
  Interventions: Device: Propel Stent
- Triamcinolone-impregnated CMC foam (Experimental): Applied to one nostril at end of case through randomization. Experimental drug is triamcinolone-acetonide 40mg/mL. 2mL will be combined with 5mL sterile water and mixed with carboxymethylcellulose foam and placed in the nares at the conclusion of the surgery. This will only be applied once and will remain in the nares until it dissolves or 7 days.
  Interventions: Drug: Triamcinolone-impregnated CMC foam

INTERVENTIONS:
Drug: Triamcinolone-impregnated CMC foam — same information as included in the arm/group descriptions
  Other Names: Kenalog-40
  Arms: Triamcinolone-impregnated CMC foam
Device: Propel Stent — same information as included in the arm/group descriptions
  Arms: Steroid-eluting implant (Propel)

SUMMARY:
This is a research study to find out if an off-label use of carboxymethylcellulose foam (CMC), an absorbable nasal packing, combined with triamcinolone acetonide, a steroid, is more comfortable postoperatively for participants and is as effective in decreasing scarring, swelling and crusting after surgery than an FDA approved steroid eluting implant. Anticipated sample size will be 30. Study is an intrapatient control design. Subjects will be randomly assigned to receive CMC foam with triamcinolone in one nare and the steroid-eluting implant in the other. Participants will fill out preoperative and follow-up visit surveys at 7, 14, 30 and 90 days. Subjects at each visit will also have pictures taken of the nasal cavities to be scored for later analysis. Paired t-tests will be performed for analysis.

Our primary objective is to demonstrate that triamcinolone-impregnated carboxymethylcellulose foam is noninferior to steroid-eluting implants in improving postoperative ethmoid inflammation, middle turbinate position, preventing intranasal synechiae and reducing polypoid change with objective measurement scales Our secondary objects include assessing the quality-of-life and nasal obstruction symptoms before and after functional endoscopic sinus surgery with validated SNOT-22 and NOSE questionnaires and to assess the cost-effectiveness of triamcinolone-impregnated carboxymethylcellulose foam versus steroid-eluting implant in management of CRSwNP in the early postoperative period.

The endpoints are the POSE scores, the SNOT-22 and NOSE scores at days 7, 14, 30 and 90.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Diagnosis of nasal polyposis and desiring surgery

Exclusion Criteria:

* A known history of intolerance to corticosteroids
* An oral steroid-dependent condition
* A history of immune deficiency
* Pre-existing narrow angle glaucoma or cataracts
* Subjects that did not complete the pre-op medical regimen described below
* Pregnant and/or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-24 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative Perioperative Sinus Endoscopy Score | 30 days
  The Perioperative Sinus Endoscopy score sums the combined scores determined from middle turbinate position, middle meatal status, ethmoid cavity appearance, as well as secondary sinus blockage (frontal and sphenoid). Each category is scored from 0-2, with 0 being not present, 1 as partially present, and 2 being fully present. The highest total score is 16, with scores ranging from 18-20 when the frontal and sphenoid sinuses are also included. The higher the score, the worse the status of the nasal cavity.
  Comparison of the mean POSE scores for the two treatments at day 30 to determine there is noninferiority

CONTACTS AND LOCATIONS:
Overall Officials: Marina Boruk, MD, Principal Investigator — SUNY Downstate Med Ctr
Locations (1):
- SUNY Downstate Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No